CLINICAL TRIAL: NCT00463853
Title: Stem Cell Therapy as Adjunct to Revascularization: STAR
Brief Title: Stem Cell Therapy as Adjunct to Revascularization
Acronym: STAR
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: inability to recruit due to administrative difficulties at the site
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLNB-017-04S
Record Dates: First submitted 2007-04-17; First posted 2007-04-20 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Coronary Arteriosclerosis; Coronary Artery Bypass Graft; Myocardial Revascularization
Keywords: Bone Marrow Cells; Cardiovascular Surgery; Coronary Artery Bypass Graft; Phase I Study; Stem Cells
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): direct intramyocardial injection of cells as adjunct to CABG
  Interventions: Procedure: Autologous stem cell therapy; Procedure: CABG; Radiation: CMRI

INTERVENTIONS:
Procedure: Autologous stem cell therapy
Procedure: CABG
Radiation: CMRI

SUMMARY:
The purpose of this study is to determine whether it is safe to receive an injection of your own bone marrow adult stem cells (autologous BM-MNC) to your heart wall during coronary artery bypass graft (CABG).

DETAILED DESCRIPTION:
The experimental design will be a Phase I safety trial in which all subjects from the VA Salt Lake City Health Care System presenting with CAD and associated depressed LV function requiring myocardial surgical revascularization will be eligible for enrollment. Patients enrolled in the study will receive autologous BM-MNC as adjunct to CABG. The primary outcome measure will be safety as measured by the incidence of postoperative Serious Adverse Events (SAE) and Adverse Events (AE). The secondary outcome measures will be LV function, myocardial perfusion, and clinical improvement. The trial will have one experiment with one patient group. Group 1 (n=15) will follow standard Phase I dose escalation curve on a magnitude of 0.5 log increase after every third patient. Dose escalation will continue until a dosage of 1 x108 cells/pt is reached or maximum tolerated dose equivalent (MTDE) is identified. Cellular therapeutic products such as BM-MNCS do not possess the same pharmacologic profile as small molecule drugs, and thus, do not possess predictable metabolic activity and metabolite production, as do traditional pharmaceuticals. This can make the identity of a maximum tolerated dose somewhat difficult. We are therefore using the term MTDE instead of MTD to indicate a cell dosage that is consistent with clinical morbidity beyond obvious clinical benefit. The characteristics identifying a MTDE could be any adverse event felt to be related to the actual cell dosage or its escalation. Although unlikely, MTDE events could include microembolic phenomena, hematoma at the injection site, obvious myocardial congestion or ischemia at the injection site.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Age 18 or older
* Ability to give informed consent
* Have documented CAD and depressed LV function (EF <40%) that is felt to be appropriately treated with surgical revascularization by the VA Salt Lake City Health Care System Cardiothoracic Surgery team and in accordance with the published 2004 ACC/AHA Guideline Update for Coronary Artery Bypass Graft Surgery; specifically, in accordance with the described indication for CABG in patients with Poor LV Function (see below).

Class I

1. CABG should be performed in patients with poor LV function who have significant left main coronary artery stenosis. (Level of Evidence: B)
2. CABG should be performed in patients with poor LV function who have left main equivalent:

   significant (greater than or equal to 70%) stenosis of the proximal LAD and proximal left circumflex artery. (Level of Evidence: B)
3. CABG should be performed in patients with poor LV function who have proximal LAD stenosis with 2- or 3-vessel disease. (Level of Evidence: B)

Class IIa

CABG may be performed in patients with poor LV function with significant viable noncontracting, revascularizable myocardium and without any of the above anatomic patterns. (Level of Evidence: B)

* NHYA/CCA Class I or higher
* Abnormal cardiac wall segment on preoperative data
* Acutely stable myocardium without evidence of cardiogenic shock or evolving myocardial infarction

Exclusion Criteria:

* EF 40%
* CAD not amenable to CABG
* ACC/AHA Poor LV Function Class III - CABG should not be performed in patients with poor LV function without evidence of intermittent ischemia and without evidence of significant revascularizable viable myocardium. (Level of Evidence: B) Evidence of intermittent ischemia is defined clinically by Cardiovascular Disease Classification (see chart above). Objectively, this can be demonstrated by various modalities that can demonstrate ischemic myocardium. Such modalities include SCA, Echo, CMRI, and radionucleotide imaging.
* Patients undergoing cardiac re-operation
* Patients with operable valvular disease
* Patients with preexisting malignant arrhythmia
* Patients with preexisting systemic malignancy
* Patients with a contraindication to MRI
* Presence of ongoing local or systemic infection
* Participation in another clinical trial
* Emergency operation
* Preoperative cardiogenic shock or evolving myocardial infarction
* ASA Class V or contraindication to general anesthesia
* Pregnancy
* Prisoner
* Active history of alcohol or substance abuse
* Active psychiatric history leading to potential for poor study participation and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be safety as measured by the incidence of postoperative serious adverse events (SAE) and adverse events (AE). | 1 year

SECONDARY OUTCOMES:
Ejection fraction measured by CMRI | at baseline, 3 & 6 months
Echo | at baseline, intervention, 2 weeks, 1 month, 3 months, 6 months and 1 year
Myocardial perfusion measured by gadolinium CMRI | at baseline, 3 & 6 months
Exercise tolerance testing | at baseline, 1 month, 3 months, 6 months, and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: G. Russell Reiss, MD, Study Chair — VA Salt Lake City Health Care System, Salt Lake City
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, Salt Lake City, Utah, United States